CLINICAL TRIAL: NCT03001622
Title: An Open Label Phase II Trial to Evaluate the Safety of IFX-1 in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Studying Complement Inhibition in Patients With Moderate to Severe Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFX-1-P2.3
Record Dates: First submitted 2016-11-29; First posted 2016-12-23 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — vilobelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFX-1 (Other)
  Interventions: Biological: IFX-1

INTERVENTIONS:
Biological: IFX-1 — chimeric, monoclonal antibody

SUMMARY:
The trial enrolls patients with moderate to severe Hidradenitis Suppurativa (HS). The primary goal of the trial is to evaluate the safety and tolerability of IFX-1 administered over 8 weeks in these patients. In addition the trial aims to characterize the pharmacokinetics and pharmacodynamics of IFX-1 as well as to generate preliminary data on the efficacy of IFX-1 on clinical endpoints (e.g., Hidradenitis Suppurativa Clinical Response (HiSCR), Dermatology Life Quality Index (DLQI), Visual Analog Scale (VAS) for disease, VAS for pain, Hidradenitis Suppurativa - Physician's Global Assessment (HS-PGA), Modified Sartorius Score (mSS)).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old
2. Written informed consent
3. Diagnosis of HS for at least 1 year
4. Hidradenitis suppurativa (HS) lesions in at least 2 distinct anatomic areas, one of which is Hurley Stage II or III
5. Total AN (abscesses and nodules) count ≥3
6. Patients with either primary or secondary failure of biological treatment or are not eligible for treatment with other biologicals
7. Failure of previous antimicrobial treatments

Exclusion Criteria:

1. Body weight above 150 kg or body weight below 60 kg
2. Has a draining fistula count of greater than 30 at baseline
3. Surgical management planned within the next 24 weeks
4. Occurrence of a flare-up of HS leading to intravenous antimicrobial treatment within the last 14 days
5. Any other disease and condition that is likely to interfere with evaluation of study product, outcome assessment or satisfactory conduct of the study

   1. Active infection
   2. Severe congestive heart failure (i.e., New York Heart Association (NYHA) Class IV)
   3. Depression
   4. History of systemic lupus erythematosus or rheumatoid arthritis
   5. Any immunodeficiency disease
   6. Active hematological or solid malignant tumor
   7. Patients must not have had any other active skin disease or condition (e.g., bacterial, fungal, or viral infection) that may have interfered with assessment of HS.
6. One of the following abnormal laboratory results

   1. White blood cell count < 2,500/mm3
   2. Neutrophil count < 1000/mm3
   3. Serum Creatinine > 3 x Upper Normal Limit (UNL)
   4. Total Bilirubin > 2 x UNL
   5. Alanine-Aminotransferase (ALAT) > 2 x UNL
   6. Positive screening test for Hepatitis B, Hepatitis C, or HIV 1/2
7. Prior administration of any biological compound in the last 3 months
8. Intake of corticosteroids defined as daily intake of prednisone or equivalent more than 1 mg/kg for the last three weeks;
9. Intake of Immunosuppressive drugs within past 30 days (e.g., cyclosporine, tacrolimus)
10. General exclusion criteria

    1. Pregnant (in women of childbearing potential an urine pregnancy test has to be performed) or breast-feeding women
    2. Women with childbearing potential (defined as within two years of their last menstruation) not willing to practice appropriate contraceptive measures (e.g., implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy, abstinence) while participating in the trial
    3. Participation in any interventional clinical trial within the last three months
    4. Known intravenous drug abuse
    5. Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least possibly related treatment-emergent adverse events (TEAEs) | up to Day 134
Number of patients with detection of anti-drug antibodies (pre-/post-dosing) | up to Day 134

SECONDARY OUTCOMES:
Plasma concentration of IFX-1 | From Day 1 until Day 134
Plasma concentration of C5a | Data will be collected at the following time points: Day 1, Day 22, Day 50 and Day 134
Percentage change from baseline in total abscess and nodule (AN) count per time point | Data will be collected at the following time points: Day 1, 22, 29, 36, 43, 50, 78, 106 and Day 134
Hidradenitis Suppurativa Clinical Response (HiSCR) per time point | Data will be collected at the following time points: Day 1, 22, 29, 36, 43, 50, 78, 106 and Day 134
Achievement of Hidradenitis Suppurativa - Physician's Global Assessment (HS-PGA) of clear, minimal, or mild among patients with at least 2 grades improvement (reduction) from baseline | Data will be collected at the following time points: Day 1, Day 22, Day 50 and Day 134
HS-PGA score per time point | Data will be collected at the following time points: Day 1, 22, 29, 36, 43, 50, 78, 106 and Day 134
Achievement of at least a 30% reduction and at least a 10 mm reduction in the Visual Analog Scale (VAS) for pain, among patients who had a baseline pain assessment ≥ 30 mm | At each visit from Day 1 until Day 134
VAS pain score per time point | At each visit from Day 1 until Day 134
Change from baseline in VAS pain score per time point | At each visit from Day 1 until Day 134
VAS disease score per time | At each visit from Day 1 until Day 134
Change from baseline in VAS disease score per time point | At each visit from Day 1 until Day 134
Dermatology Life Quality Index (DLQI) per time point | Data will be collected at the following time points: Day 1, Day 22, Day 50 and Day 134
Change from baseline in DLQI per time point | Data will be collected at the following time points: Day 1, Day 22, Day 50 and Day 134

CONTACTS AND LOCATIONS:
Locations (1):
- ATTIKON University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prens LM, Ardon CB, van Straalen KR, van der Zee HH, Seelen MAJ, Laman JD, Prens EP, Horvath B, Damman J. No Evident Systemic Terminal Complement Pathway Activation in Hidradenitis Suppurativa. J Invest Dermatol. 2021 Dec;141(12):2966-2969.e1. doi: 10.1016/j.jid.2021.03.037. Epub 2021 Jul 9. No abstract available. PMID 34252397